CLINICAL TRIAL: NCT02204722
Title: A Phase IV Study to Evaluate Efficacy and Safety of Imatinib(Glinib®) 600mg/Day Depending on Early Molecular Response in Newly Diagnosed Patients With Chronic Myeloid Leukemia in Chronic Phase
Brief Title: A Study to Evaluate Efficacy and Safety of Glinib in Newly Diagnosed CML Patients
Acronym: IDEAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's decision to halt the study.
Sponsor: Dong-A ST Co., Ltd. (Industry)
Collaborators: SeoulCRO (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA_CML_IV
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B (Experimental): the group who has more than 10% of the BCR-ABL(IS) level for three months will receive 600mg/day of Imatinib after three months.
  Interventions: Drug: 600mg/day of Imatinib
- Group A (Experimental): the group who has more than 10% of the BCR-ABL(IS) level for three months will maintain the dose, 400mg/day of Imatinib, after three months.
  Interventions: Drug: 400mg/day of Imatinib

INTERVENTIONS:
Drug: 600mg/day of Imatinib
  Arms: Group B
Drug: 400mg/day of Imatinib
  Arms: Group A

SUMMARY:
This study is to evaluate efficacy and safety of Imatinib in two groups of patients; all patients should be diagnosed less than 3 months as chronic myeloid leukemia in a chronic phase. The group A, the reference group, will have 10% or less than 10% of the BCR-ABL level after three month dosing and be maintained their dose of 400mg/day. On the other hand, the group B, will have more than 10% and the dose will be increased from 400mg/day to 600mg/day. The superiority of the group B will be proved by evaluating the MMR rate of these two groups after 12 months of administeration of Imatinib.

ELIGIBILITY:
Inclusion Criteria:

* at the age of 18 or more
* newly diagnosed within three months as a Chronic Myeloid Leukemia
* with positive Philadelphia chromosome and appearance of BCR-ABL transcript
* with 0 - 2 of ECOG Performance Status
* with normal renal function
* with normal hepatic function
* able to understand and decide to involve the study

Exclusion Criteria:

* history of radiation therapy for more than 25% of bone marrow due to other malignant diseases
* history of other clinically relevant malignant tumors
* with bleeding disorders which are not related to leukemia
* evidence of clinically relevant cardiac dysfunction
* with severe disease which cannot be regulated by other organs
* a previous administration of Imatinib more than a week prior to the first dose.
* participation in other drug study(eg. intervention trial) within 30 days prior to the screening visit
* HIV-infected
* females with pregnancy, childbearing or lactating potential
* other reasons determined by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
MMR rate at 12 months in two groups | 12 months
  MMR rate at 12 months in two groups will be compared. Group A is consisted of patients with equal or less than 10% of BDR-ABL, Group B is consisted of patients with more than 10% of BDR-ABL.

SECONDARY OUTCOMES:
CCyR in group A and B | 12 months
  CCyR rate for 12 months and the duration of the complete CCyR will be evaluated.
MMR in group A and B | 12 months
  MMR rate for 12 months and the duration of MMR will be measured.
CMR in group A and B | 12 months
Survival rate in group A and B | 12 months
Progression rate to AP/BC in group A and B | 12 months
the actual administration | 12 months
  the total dose will be divided by total days of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Hyoung Lee, M.D., Principal Investigator — Asan Medical Center; Jin-hee Park, M.D., Principal Investigator — Gachon University Gil Medical Center; Chul-won Choi, M.D., Principal Investigator — Korea University Guro Hospital; Sae-ryun Lee, M.D., Principal Investigator — Korea University Ansan Hospital; Yong Park, M.D., Principal Investigator — Korea University Anam Hospital; Joo-sup Joeng, M.D., Principal Investigator — Pusan National University Hospital; Jung-ok Lee, M.D., Principal Investigator — Seoul National University Bundang Hospital; Chul-won Jung, M.D., Principal Investigator — Seoul Medical Center; Sung-soo Yoon, M.D., Principal Investigator — Seoul National University Hospital; Kyung-ha Kim, M.D., Principal Investigator — Soonchunhyang University Hospital Seoul; Joon-sung Park, M.D., Principal Investigator — Ajou University School of Medicine; Duk-yeon Cho, M.D., Principal Investigator — Chungnam National University Hospital; Sung-nam Im, M.D., Principal Investigator — Inje University Haeundae Paik Hospital
Locations (1):
- Asan Medical Center, Seoul, South Korea